CLINICAL TRIAL: NCT02855125
Title: A Randomized, Open-Label, Multi-Center, International Phase 2 Study of TAS-114 in Combination With S-1 in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Randomized Phase 2 Trial of TAS-114 in Combination With S-1 Versus S-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-114-201; 2016-001806-40 (EudraCT Number)
Record Dates: First submitted 2016-07-18; First posted 2016-08-04 (Estimated); Results first posted 2021-12-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: NSCLC; phase 2 study; TAS-114; S-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TAS-114; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAS-114 + S-1 (Active Comparator): Participants received 400 milligrams (mg) of TAS-114 tablets orally twice daily (BID) along with 30 milligrams per meter square (mg/m^2) of S-1 capsule BID for 2 weeks (Day 1 to 14), followed by 1 week recovery period (Day 15 to 21) in each 21 days cycle, until progressive disease (PD), occurrence of intolerable side effects, removal by the Investigator, or withdrawal of consent (maximum treatment duration: 51 weeks).
  Interventions: Drug: TAS-114; Drug: S-1
- S-1 (Monotherapy) (Active Comparator): Participants received 30 mg/m^2 of S-1 capsules BID for 2 weeks (Day 1 to 14) followed by 1 week recovery period (Day 15 to 21) in each 21 days cycle, until progressive disease (PD), occurrence of intolerable side effects, removal by the Investigator, or withdrawal of consent (maximum treatment duration: 38 weeks).
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: TAS-114 — TAS-114 was a modulator of 5-fluorouracil (5-FU).
  Arms: TAS-114 + S-1
Drug: S-1 — S-1 was designed to provide oral delivery of 5-FU and to reduce the rate of degradation of 5-FU in vivo.

SUMMARY:
This is a randomized, open-label, Phase 2 study of TAS-114 administered in combination with S-1, to investigate the efficacy, safety and tolerability of the TAS-114/S-1 regimen in patients with advanced or metastatic NSCLC.

The study will be conducted internationally in 2 regions: Asian [Japan] and Western [Europe and US]. Patients will be randomized into TAS-114/S-1 arm versus S-1 control arm in a 1:1 ratio.

DETAILED DESCRIPTION:
Randomization will take place once the consented patient has completed all the necessary baseline procedures and is deemed eligible for study entry. Treatment assignment will be done centrally using a dynamic allocation method (biased coin) via an interactive voice/web response system (IXRS) stratified by:

* Geographical region (Region 1: Asian [Japan]; Region 2: Western [Europe and US])
* Histological subtypes (nonsquamous cell carcinoma [including mixed] and squamous cell carcinoma)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old (≥ 20 years old in Japan);
2. Histologically diagnosed or cytologically proven advanced or metastatic NSCLC patients, either Stage IIIB/Stage IV disease (according to Version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology), or recurrent disease following radiation therapy or surgical resection;
3. Patients who had received at least 2 prior therapies for advanced or metastatic disease condition, including platinum doublet and pemetrexed, docetaxel, or immunotherapy, and were refractory to or unable to tolerate their last prior therapy
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Version 1.1, 2009);
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
6. Predicted life expectancy of at least 3 months;
7. Able to take medications orally;
8. Adequate organ function
9. Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum) within 7 days prior to starting the study drug. Both males and females must agree to use effective birth control during the study (prior to the first dose and for 6 months after the last dose) if conception is possible during this interval.
10. Willing and able to comply with required scheduled visits and study procedures.

Exclusion Criteria:

1. Treatment with any of the following within the specified time frame prior to the study drug administration:

   * Major surgery within prior 4 weeks and minor surgery within 7 days;
   * Radiotherapy for extended field within prior 4 weeks or limited field within prior 2 weeks;
   * Any anticancer therapy or investigational agent within prior 3 weeks.
2. A serious illness or medical condition
3. Concomitant treatment with the following drugs that may interact with S-1:

   Sorivudine, brivudine, uracil, eniluracil, folinate/folinic acid, Cimetidine, dipyridamole, and nitroimidazoles, including metronidazole and misonidazoleMethotrexate, Clozapine,Allopurinol,Phenytoin,Flucytosine, a fluorinated pyrimidine antifungal agent,Coumarin-derivative anticoagulant
4. Known hypersensitivity to S-1 or its metabolites (eg, 5-FU);
5. Previous use of TAS-114, S-1, and 5-FU drugs;
6. A pregnant or lactating female or possibly pregnant women, or men or women wishing to have children during the study period;
7. A judgment of the investigator that the patient is inappropriate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Central, Study Director — Taiho Oncology, Inc. USA
Locations (30):
- United States (6):
  - Loma Linda, California
  - Gainesville, Florida
  - Cleveland, Ohio
  - Portland, Oregon
  - Dallas, Texas
  - Seattle, Washington
- France (6):
  - Caen
  - Lille
  - Marseille
  - Paris
  - Pierre-Bénite
  - Villejuif
- Italy (4):
  - Catania
  - Milan
  - Palermo
  - Ravenna
- Japan (7):
  - Kashiwa, Chiba
  - Sayama, Osaka
  - Adachi, Saitama
  - Chuo-Ku, Tokyo
  - Koto-Ku, Tokyo
  - Sunto-Gun, Tokyo
  - Wakayama
- Poland (4):
  - Katowice
  - Lodz
  - Lublin
  - Warsaw
- Spain (3):
  - Badalona
  - Barcelona
  - Madrid

REFERENCES:
- [Derived] Yamamoto N, Hayashi H, Planchard D, Moran T, Gregorc V, Dowell J, Sakai H, Yoh K, Nishio M, Cortot AB, Benhadji KA, Soni N, Huang J, Makris L, Cedres S. A randomized, phase 2 study of deoxyuridine triphosphatase inhibitor, TAS-114, in combination with S-1 versus S-1 alone in patients with advanced non-small-cell lung cancer. Invest New Drugs. 2020 Oct;38(5):1588-1597. doi: 10.1007/s10637-020-00930-5. Epub 2020 Apr 3. PMID 32246224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 centers in 5 countries.
Pre-assignment Details: A total of 128 participants were randomized.1 participant in S-1 (Monotherapy) arm was randomized but not treated.
Period: Overall Study
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Started | 64 | 64
Treated | 64 | 63
Completed | 0 | 0
Not Completed | 64 | 64
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Clinical Disease Progression | 5 | 4
Not completed — Radiologic Disease Progression | 36 | 39
Not completed — Adverse Event | 11 | 7
Not completed — Physician Decision | 1 | 0
Not completed — On Treatment | 9 | 11
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included all participants randomized in the study, regardless of whether they actually received any study treatment (TAS-114 or S-1) or not.
Groups:
- TAS-114 + S-1: Participants received 400 mg of TAS-114 tablets orally BID along with 30 mg/m^2 of S-1 capsule BID for 2 weeks (Day 1 to 14), followed by 1 week recovery period (Day 15 to 21) in each 21 days cycle, until progressive disease (PD), occurrence of intolerable side effects, removal by the Investigator, or withdrawal of consent (maximum treatment duration: 51 weeks).
- Total: Total of all reporting groups
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy) | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (7.77) | 62.6 (10.22) | 63.2 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 41 | 48 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 45 | 47 | 92
  Unknown or Not Reported | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Central Independent Review
Description: Progression-free survival was defined as the time (in months) from the day of randomization to the start of radiologic disease progression or death (any cause), whichever occurred first. Response assessments were made based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). As per RECIST 1.1 criteria, progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). (Note: the appearance of one or more new lesions was also considered progressions). Participants who did not have disease progression or died were censored at the last known time that the participant was progression free.
Time Frame: From date of randomization or until date of disease progression or death whichever occurred first (approximately up to 13 months)
Population: Intent-to-Treat (ITT) population included all participants randomized in the study, regardless of whether they actually received any study treatment (TAS-114 or S-1) or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Number analyzed (Participants) | 64 | 64
months | 3.65 [2.69 to 5.16] | 4.17 [2.60 to 6.60]
Statistical Analysis 1: Comparison: TAS-114 + S-1 vs S-1 (Monotherapy); Test type: Superiority; p = 0.2744, Log Rank; 1-sided stratified log-rank test; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.71 to 1.88] — Based on stratified Cox regression model

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of the study treatment to death from any cause. Participants who were alive at the end of study were censored at the last date the participant was known to be alive. OS was estimated from Kaplan-Meier method.
Time Frame: From date of randomization until death (approximately up to 15 months)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Number analyzed (Participants) | 64 | 64
months | 7.92 [6.28 to 10.78] | 9.82 [7.66 to 13.40]
Statistical Analysis 1: Comparison: TAS-114 + S-1 vs S-1 (Monotherapy); Test type: Superiority; p = 0.1431, Log Rank; 1-sided stratified log-rank test; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.80 to 2.14] — Based on stratified Cox regression model

3. Secondary Outcome: Overall Response Rate (ORR) Based on Central Independent Review
Description: ORR was defined as the percentage of participants with objective evidence of complete response (CR) or partial response (PR) per response evaluation criteria in solid tumors (RECIST) version 1.1. CR was defined as the disappearance of all target lesions and non-target lesions and normalization of tumor marker level. Any pathological and non-pathological lymph nodes must have reduction in short axis to less than (<) 10 mm. PR was defined as at least a 30 percent (%) decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters.
Time Frame: From date of first dose of study drug to the date of first documentation of progression or death (approximately up to 13 months)
Population: Tumor response (TR) population included all participants randomized in the study, regardless of whether they actually received any study treatment (TAS-114 or S-1) or not; with measurable disease (at least one target lesion) at baseline and with at least one tumor evaluation (participants who had disease progression or had a cancer related death prior to their 1st tumor evaluation were also considered evaluable).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Number analyzed (Participants) | 61 | 58
percentage of participants | 19.7 [10.6 to 31.8] | 10.3 [3.9 to 21.2]

4. Secondary Outcome: Disease Control Rate (DCR) Based on Central Independent Review
Description: DCR was defined as the percentage of participants with objective evidence CR, PR, or stable disease (SD). Based on the central review of tumor assessments per RECIST, version 1.1. CR was defined as disappearance of all target lesions. Reduction in any pathological lymph nodes in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as a reference the smallest sum diameters during study.
Time Frame: as for outcome 3
Population: TR population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Number analyzed (Participants) | 61 | 58
percentage of participants | 80.3 [68.2 to 89.4] | 75.9 [62.8 to 86.1]

5. Secondary Outcome: Duration of Response (DR) Based on Central Independent Review
Description: DR was derived for participants with objective evidence of PR or CR. DR was defined as the time (in months) from the first documentation of response (CR or PR) to the first documentation of objective tumor progression or death due to any cause. Participants who were alive and progression-free as of the analysis cut-off date were censored at their last evaluable tumor response assessment before initiation of any new anticancer treatment.
Time Frame: From date of first response to the date of first documentation of progression or death (approximately up to 13 months)
Population: TR population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Number analyzed (Participants) | 12 | 6
months | 3.38 [2.37 to 4.86] | NA [2.79 to NA] — Median and upper limit of 95% Confidence interval were not estimable because of censoring in 5 of the 6 participants.

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical condition that occurs in a participants while participating in a clinical study and does not necessarily have a causal relationship with the use of the study treatment. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as AEs that developed or worsened during the TEAE period which was defined as the period from the time of first dose of study treatment until 30 days after last dose of study treatment. AEs included both serious and non- serious adverse events.
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (approximately up to 13 months)
Population: Analysis was performed on As-Treated (AT) population which included all participants who received at least 1 dose of TAS-114 or S-1.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
Number analyzed (Participants) | 64 | 63
Participants
  Participants with TEAEs | 64 | 61
  Participants with TESAEs | 30 | 19

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (approximately up to 13 months)
Description: Analysis was performed on As-Treated (AT) population which included all participants who received at least 1 dose of TAS-114 or S-1.
Arm/Group | TAS-114 + S-1 | S-1 (Monotherapy)
All-Cause Mortality (participants affected / at risk) | 36/64 | 29/63
Serious Adverse Events (participants affected / at risk) | 30/64 | 19/63
Other Adverse Events (participants affected / at risk) | 64/64 | 61/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-114 + S-1 (N=64) | S-1 (Monotherapy) (N=63)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1)
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Disease progression (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-114 + S-1 (N=64) | S-1 (Monotherapy) (N=63)
Anaemia (Blood and lymphatic system disorders) | 42 (111) | 17 (26)
Neutropenia (Blood and lymphatic system disorders) | 5 (14) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 2 (5)
Lacrimation increased (Eye disorders) | 5 (5) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 3 (6)
Constipation (Gastrointestinal disorders) | 9 (9) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 19 (32) | 18 (24)
Nausea (Gastrointestinal disorders) | 20 (61) | 23 (62)
Stomatitis (Gastrointestinal disorders) | 10 (18) | 4 (5)
Vomiting (Gastrointestinal disorders) | 12 (32) | 13 (18)
Asthenia (General disorders) | 19 (40) | 14 (22)
Fatigue (General disorders) | 6 (12) | 11 (18)
Malaise (General disorders) | 10 (18) | 5 (6)
Mucosal inflammation (General disorders) | 4 (5) | 3 (3)
Non-cardiac chest pain (General disorders) | 6 (7) | 3 (4)
Oedema peripheral (General disorders) | 5 (6) | 4 (7)
Pyrexia (General disorders) | 14 (17) | 9 (12)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5)
Alanine aminotransferase increased (Investigations) | 3 (7) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 6 (9)
Blood bilirubin increased (Investigations) | 0 (0) | 5 (12)
Lymphocyte count decreased (Investigations) | 4 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (25) | 7 (11)
Platelet count decreased (Investigations) | 8 (18) | 6 (11)
Weight decreased (Investigations) | 5 (6) | 0 (0)
White blood cell count decreased (Investigations) | 10 (34) | 5 (10)
Decreased appetite (Metabolism and nutrition disorders) | 29 (46) | 27 (44)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (13) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 4 (6)
Headache (Nervous system disorders) | 4 (6) | 3 (4)
Insomnia (Psychiatric disorders) | 5 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 7 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 10 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (14) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (13) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 15 (29) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (46) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 18 (25) | 12 (12)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT02855125/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT02855125/SAP_001.pdf